CLINICAL TRIAL: NCT00088374
Title: A Phase II Study of 17-Allylamino-17-Demethoxygeldanamycin in Patients With Von Hippel Lindau Disease and Renal Tumors
Brief Title: 17AAG to Treat Kidney Tumors in Von Hippel-Lindau Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: William M. Linehan, M.D., National Cancer Institute, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 040238; 04-C-0238 (Other: Clinical Center (CC), National Institutes of Health (NIH)); 040238 (Other: Clinical Center (CC), National Institutes of HEalth (NIH)); NCT00089375 (obsolete NCT alias)
Record Dates: First submitted 2004-07-23; First posted 2004-07-26 (Estimated); Results first posted 2011-09-29 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: Hippel-Lindau Disease; Kidney Cancer
Keywords: Kidney Cancer; VHL; 17 AAG; Chemotherapy; Von Hippel Lindau Disease; Renal Tumor
MeSH Terms: conditions — von Hippel-Lindau Disease; Kidney Neoplasms; Carcinoma, Renal Cell | interventions — tanespimycin; Fluorodeoxyglucose F18; Oxygen-15

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Von Hippel-Lindau (VHL) associated renal tumors (Experimental)
  Interventions: Drug: 17 allylamino-17-demethoxygeldanamycin; Drug: 18 FDG (Fludeoxyglucose 18F); Drug: [15-O] H2O; Drug: EPL diluent

INTERVENTIONS:
Drug: 17 allylamino-17-demethoxygeldanamycin — 17 allylamino-17-demethoxygeldanamycin (17 AAG) given intravenously at a dose of 300 mg/m2 on days 1,8 and 15 of 28 day cycles.
  Other Names: 17 AAG
Drug: 18 FDG (Fludeoxyglucose 18F) — 18FDG PET performed at baseline and 12 weeks after treatment. At each timepoint participants can receive 250mCi 0-15 water and 15 mCi F18-FDG.
  Other Names: Fludeoxyglucose (18F)
Drug: [15-O] H2O — [15-0] H20 performed at baseline and 12 weeks after treatment. At each time point participants can receive 250mCi 0-15 water and 15 mCi F18-FDG. The water scans were done as several intravenous injections for several scans but not over a total of 250 mCi.
  Other Names: water scan
Drug: EPL diluent — 17AAG is formulated with this diluent. Supplied in a 50 mL flint vial containing 48 mL of 2% egg phospholipids, and 5% dextrose in Water for Injection, USP. Patients with a history of serious allergic reactions to eggs should not receive this agent.
  Other Names: Egg phospholipid

SUMMARY:
This study will examine whether the drug 17AAG (17-allylamino 17-demethoxygeldanamycin) can shrink kidney tumors in patients with Von Hippel-Lindau disease (VHL), a rare, inherited syndrome in which patients develop tumors in certain parts of the body. 17AAG contributes to the destruction of proteins in cells that may play in role in causing cancer and spurring tumor growth. The study will also look at the effect of 17AAG on other tumors patients may have that are caused by VHL, on the amount of blood vessels in the tumors, on the biologic activity of the tumor, and on cells circulating in the bloodstream, as well as the safety of the drug and its impact on the kidney tumor in patients whose tumor(s) is removed.

Patients 18 years of age and older with von Hippel-Lindau disease who have at least one kidney tumor large enough to pose a risk of metastasis (spread of cancer to other parts of the body) may be eligible for this study. Candidates are screened with a medical history and physical examination, computed tomography (CT) scan, brain magnetic resonance imaging (MRI), see below), and blood and urine tests. Additional tests, including a 24-hour urine collection, ultrasound of the testicles in men, hearing test, eye exam, and MRI of the spine, may be done if recent test results are not available.

Participants undergo the following tests and procedures:

MRI: This test uses a strong magnetic field and radio waves to show structural and chemical changes in tissue. During the scan, the patient lies on a table in a narrow cylinder containing a magnetic field, wearing earplugs to muffle loud noises that occur with electrical switching of the magnetic fields. A catheter (plastic tube) is inserted into the patient's arm to administer a contrast dye that enhances the images.

17AAG treatment: Patients receive 17AAG infusions into a vein once a week for 3 weeks out of every 4, for 3 months. The infusions last up to 1 to 2 hours.

Repeat testing: After 3 months, patients have repeat MRI scans to measure changes in tumor activity, blood flow, and number of blood vessels in the tumor since the pretreatment scans. They may have additional tests, including a CT scan, eye exam, and other tests to evaluate the effect of 17AAG on the tumors.

DETAILED DESCRIPTION:
Background:

Von Hippel-Lindau disease is a hereditary cancer syndrome in which affected individuals are at risk for developing tumors in a number of organs, including the brain, spine, adrenal glands, eyes and pancreas.

The molecular hallmark of VHL is inactivation of the VHL gene which leads to accumulation of the hypoxia inducible factors (HIF); this, in turn results in overexpression of several genes including vascular endothelial growth factor (VEGF), glucose transporter 1 (GLUT-1), transforming growth factor alpha (TGF-α), platelet-derived growth factor (PDGF) and erythropoietin, which play an important role in tumorigenesis, tumor growth and metastasis.

17-allylamino-17-demethoxygeldanamycin (17AAG) is an inhibitor of the cellular chaperone heat shock protein 90 (Hsp90), and its interaction with Hsp90 leads to destabilization and degradation of several proteins, that depend on Hsp90 for their stability.

The alpha subunit of HIF1 is one such Hsp90 client protein' and is susceptible to VHL independent, 17AAG-induced degradation.

Objectives:

To evaluate the efficacy of 17 AAG administered as a single agent in von Hippel Lindau patients with renal tumors. The primary endpoint of the trial is response of renal tumors following 3 cycles of therapy.

To study the safety and tolerability of 17 AAG. To evaluate PD modulation of hsp90, and to explore the utility dynamic contrast enhanced MRI in evaluation of blood flow and metabolic changes in renal tumors before and during therapy

Eligibility:

Adults with clinical diagnosis of von Hippel Lindau disease Presence of one or more localized renal tumors for which surgical resection would be considered the standard approach

Design:

Patients will receive 17 AAG as an intravenous infusion at a dose of 300mg/m(2) on days 1, 8, and 15 of 28 day cycles.

The study will follow a two-stage MinMax phase II design and will accrue a maximum of 26 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must satisfy all of the following inclusion criteria to be eligible for study enrollment.
* Clinical diagnosis of von Hippel Lindau disease.
* Presence of one or more localized renal tumors for which surgical resection would be considered the standard approach.
* Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of 17 AAG in patients less than 18 years of age, children are excluded from this study.
* Life expectancy less than 3 months.
* Performance status Eastern Cooperative Oncology Group (ECOG) 0-2.
* Patients must have normal organ and marrow function as defined below: white blood cells (WBC)count greater than or equal to 3,000/microliter, absolute neutrophil count greater than or equal to 1,500/microliter, platelet count greater than or equal to 100,000/microliter, Hgb greater than 10Gm/dl, serum creatinine less than or equal to 1.0 upper limit of normal (ULN) or measured 24 hour creatinine clearance greater than 60 ml/min,aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than 1.0 times the ULN, total bilirubin less than or equal to ULN(less than 3 times the normal limit (NL) in patients with Gilbert's disease).
* Negative hepatitis B surface antigen (HbsAg), human immunodeficiency virus type 1 (HIV-1) and nonreactive hepatitis C virus (HCV).
* No history of serious intercurrent illness.
* At least four weeks from completion of any surgical or investigational therapy for von Hippel Lindau disease.
* Willingness to undergo resection of renal tumor at the time point defined in the protocol.
* All men and women of childbearing potential must use effective contraception as determined by the principal investigator or protocol chair.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior or concomitant non-von Hippel Lindau associated malignancy with the exception of adequately treated basal or squamous cell carcinoma of the skin or any other malignancy from which the patient has remained disease free for more than five years.
* Any renal tumor greater than 4cm in size.
* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events (to grade 1 or less toxicity according to Common Terminology Criteria for Adverse Events version 3.0 (CTCAE 3.0) due to agents administered more than 4 weeks earlier.
* Patients may not be receiving any other investigational agents.
* Patients with known metastatic renal cell cancer.
* Patients with a history of serious allergy to eggs.
* Concomitant therapy with cytochrome P450 3A4 (CYP3A4) potent inhibitors.
* Patients who are on CYP3A4 substrates and inducers qualify for enrollment for this study.
* Pregnant women are excluded from this study because 17 AAG has the potential for teratogenic or abortifacient effects, and no data regarding its safety in pregnant women is available. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with 17 AAG, breastfeeding should be discontinued if the mother is treated with 17 AAG.
* Human immunodeficiency virus (HIV)-positive patients are excluded from the study because of unknown but potential pharmacokinetic interactions of anti-retroviral drugs with 17 AAG.
* Use of any medications that prolong or may prolong corrected QT interval (QTc).
* Patients who have significant cardiac disease including heart failure that meets New York Heart Association (NYHA)class III and IV definitions, uncontrolled dysrhythmias requiring anti-arhythmic drugs, or patients with active ischemic heart disease including myocardial infarction and poorly controlled angina within 12 months of study entry.
* Patients who have a history of serious ventricular arrhythmia (ventricular tachycardia (VT) or ventricular fibrillation (VF),greater than or equal to 3 beats in a row), QTc greater than or equal to 450msec for men and 470msec for women, or left ventricular ejection fraction (LVEF) below lower limit of normal by multi gated acquisition scan(MUGA).
* Patients with a history of prior chest radiation or radiation that potentially included the heart in the treatment field.
* Patients with congenital long Q wave, T wave (QT) syndrome.
* Patients with left bundle branch block.
* Patients with symptomatic pulmonary disease requiring medication, including the following:dyspnea, dyspnea on exertion, paroxysmal nocturnal dyspnea, oxygen requirement and significant pulmonary disease, including chronic obstructive pulmonary disease, patients meeting Medicare criteria for home oxygen.
* Carbon monoxide diffusing capacity (DLCO) less than or equal to 80%.
* Patients with a prior history of cardiac or pulmonary toxicity after receiving anthracyclines, such as doxorubicin, daunorubicin, mitoxantrone, bleomycin, or carmustine (BCNU).
* Patients with greater than or equal to grade 2 baseline pulmonary or cardiac symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2004-07; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William M Linehan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute, National Institutes of Health, Bethesda, Maryland, United States

REFERENCES:
- [Background] Linehan WM, Lerman MI, Zbar B. Identification of the von Hippel-Lindau (VHL) gene. Its role in renal cancer. JAMA. 1995 Feb 15;273(7):564-70. No abstract available. PMID 7837390
- [Background] Clifford SC, Maher ER. Von Hippel-Lindau disease: clinical and molecular perspectives. Adv Cancer Res. 2001;82:85-105. doi: 10.1016/s0065-230x(01)82003-0. PMID 11447766
- [Background] Maher ER, Kaelin WG Jr. von Hippel-Lindau disease. Medicine (Baltimore). 1997 Nov;76(6):381-91. doi: 10.1097/00005792-199711000-00001. PMID 9413424
- See also: Genetics Home Reference — http://ghr.nlm.nih.gov
- See also: Medline Plus — http://www.nlm.nih.gov/medlineplus/
- See also: Drug Information — http://druginfo.nlm.nih.gov/drugportal/drugportal.jsp
- See also: U.S FDA Resources — http://www.clinicaltrials.gov/ct2/info/fdalinks
- See also: Revised RECIST guideline version 1.1 — http://ctep.cancer.gov/protocol/Development/docs/recist_guideline.pdf
- See also: NCI Common Terminology Criteria for Adverse Events — http://ctep.cancer.gov/reporting/ctc.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The accrual ceiling for this study is 25 patients. With an expected accrual of 10-12 patients per year, we expect to complete the accrual within 2-3 years.
Groups:
- VHL Associated Renal Tumors: 17-AAG intravenous infusions at a dose of 300 mg/m2 into a vein once a week for 3 weeks out of every 4, for 3 months; on days 1, 8, and 15 of 28 cycles. The infusions last up to 1 to 2 hours.
Period: Overall Study
Arm/Group | VHL Associated Renal Tumors
Started | 9
Completed | 7
Not Completed | 2
Not completed — patient did not receive any 17AAG | 1
Not completed — patient received <1 cycle only of 17AAG | 1

BASELINE CHARACTERISTICS:
Arm/Group | VHL Associated Renal Tumors
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 48.32 (10.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Renal Tumor Response
Description: Response is defined as the number of patients who experience a disease response (complete response (CR) or partial response (PR) of renal tumors)per RECIST criteria. CR is the disappearance of all target lesions. PR is at least a 20% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. See the protocol Link module for the full criteria if desired.
Time Frame: 12 weeks
Population: 8 patients were evaluable (received at least one dose of drug and had a follow up scan).
Measure: Number; unit: participants
Arm/Group | Participants With VHL Associated Renal Tumors
Number analyzed (Participants) | 8
participants | 0

2. Secondary Outcome: Number of Participants With a Non-renal Tumor Response
Description: Number of patients who have a PR or CR of non-renal lesions (pancreatic tumors, pheochromocytomas, and hemangioblastomas). The effect of treatment on the lesions will be evaluated at baseline and at the time of restaging (12 weeks) per RECIST criteria. RECIST is defined as changes in only the largest diameter (unidimensional measurement) of the tumor lesions. Lesions are either measurable or non-measurable using the criteria. See the protocol Link module for the full criteria if desired.
Time Frame: Baseline and 12 weeks
Population: There were only two patients with measurable nonrenal tumors and hence the number of participants analyzed is correct.
Measure: Number; unit: participants
Arm/Group | Participants With VHL Associated Renal Tumors
Number analyzed (Participants) | 2
participants | 0

3. Secondary Outcome: The Number of Participants With Adverse Events
Description: Here are the total number of participants with adverse events. For the detailed list of adverse events see the adverse event module.
  The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 will be utilized for adverse event reporting. For a detailed description see the link in the Protocol Link module.
Time Frame: 1 yr, 364 days
Measure: Number; unit: participants
Arm/Group | Participants With VHL Associated Renal Tumors
Number analyzed (Participants) | 9
participants | 9

4. Secondary Outcome: The Number of Participants With HIF, HSP90, and HSP70 Modulation in Resected Tumor Tissue and/or Peripheral Blood Lymphocytes
Description: Measurement of HIF, HSP90 and HSP70 levels by Western Blot in tumor tissue and/or lymphocytes to assess modulation of these biomarkers in response to 17 AAG treatment. Pretreatment tumor samples (when available) and resected tumors (in those patients who did not have a response and underwent surgical resection of their tumor) were to be used for this analysis. Levels of Hsp90, Hsp70, HIF and HIF transcriptional targets in resected tumor will be compared to respective levels in tumors previously resected from other VHL patients (not treated with 17AAG).
Time Frame: Baseline and 12 weeks
Population: This analysis was not performed as it was felt that there were not a sufficient number of samples to enable a meaningful analysis.
Arm/Group | Participants With VHL Associated Renal Tumors
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Patients in Whom Renal Tumors Could be Identified by Positron Emission Tomography (PET)Based on Fludeoxyglucose 18F (18FDG) Uptake
Description: Images were acquired after the intravenous administration of 18FDG and H2015 and used to analyze glucose uptake and estimate blood flow. The parameter to be measured is SUV (standard uptake value(s)) and/or mL/min/gm.
Time Frame: Baseline and at 12 weeks
Population: Response was not the endpoint. The SUV values were in the 2-3 range and hence renal tumors could not be clearly identified by this technique in any of the patients.
Measure: Number; unit: participants
Arm/Group | Participants With VHL Associated Renal Tumors
Number analyzed (Participants) | 5
participants | 0

6. Secondary Outcome: Number of Participants With Flow Dynamics Measured by DCE MRI Within the Renal and Non-renal Tumor
Description: Dynamic images will be acquired before and after the intravenous administration of 0.1 mmol/kg of Gadolinium Diethylene triamine pentaacetic acid (DTPA). Time activity curves will be generated over a period of ten minutes. The parameter to be measured is the forward contrast transfer rate (Ktrans), the reverse contrast transfer rate (Kep), and/or the extravascular extracellular space volume fraction (Ve). Flow dynamics are a measure of blood flow changes in the tumor and are determined using the parameters we had previously defined (Ktrans, Kep, etc.).
Time Frame: Baseline and during therapy (12 weeks)
Population: It is not the magnitude of changes in Ktrans, Kep, and Ve that limit our abililty, but the fact that this data was available in only a small number of patients.
Measure: Number; unit: participants with changes
Arm/Group | Participants With VHL Associated Renal Tumors
Number analyzed (Participants) | 4
participants with changes | 3

ADVERSE EVENTS:
Time Frame: 2 years, 364 days
Arm/Group | Participants With VHL Associated Renal Tumors
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With VHL Associated Renal Tumors (N=9)
Dizziness (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With VHL Associated Renal Tumors (N=9)
ALLERGY/IMMUNOLOGY:: Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 3 (3)
BLOOD/BONE MARROW:: Hemoglobin (Investigations) | 1 (1)
BLOOD/BONE MARROW:: Leukocytes (total WBC) (Investigations) | 1 (2)
BLOOD/BONE MARROW:: Lymphopenia (Investigations) | 1 (2)
CARDIAC ARRHYTHMIA:: Conduction abnormality/atrioventricular heart block:: AV Block-First degree (Cardiac disorders) | 1 (5)
CARDIAC ARRHYTHMIA:: Conduction abnormality/atrioventricular heart block:: AV Block-Second degree Mo (Cardiac disorders) | 1 (1)
CARDIAC ARRHYTHMIA:: Palpitations (Congenital, familial and genetic disorders) | 1 (1)
CARDIAC ARRHYTHMIA:: Supraventricular and nodal arrhythmia:: Sinus bradycardia (Cardiac disorders) | 3 (14)
CARDIAC ARRHYTHMIA:: Supraventricular and nodal arrhythmia:: Sinus tachycardia (Cardiac disorders) | 1 (1)
CARDIAC ARRHYTHMIA:: Ventricular arrhythmia:: Ventricular tachycardia (Cardiac disorders) | 1 (2)
CARDIAC GENERAL:: Left ventricular diastolic dysfunction (Cardiac disorders) | 1 (1)
CONSTITUTIONAL SYMPTOMS:: Fatigue (asthenia, lethargy, malaise) (General disorders) | 5 (14)
CONSTITUTIONAL SYMPTOMS:: Insomnia (General disorders) | 2 (2)
CONSTITUTIONAL SYMPTOMS:: Odor (patient odor) (General disorders) | 1 (1)
CONSTITUTIONAL SYMPTOMS:: Weight gain (General disorders) | 1 (1)
CONSTITUTIONAL SYMPTOMS:: Weight loss (General disorders) | 1 (2)
DERMATOLOGY/SKIN:: Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
DERMATOLOGY/SKIN:: Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 (2)
GASTROINTESTINAL:: Anorexia (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL:: Constipation (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL:: Diarrhea (Gastrointestinal disorders) | 2 (5)
GASTROINTESTINAL:: Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL:: Heartburn/dyspepsia (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL:: Nausea (Gastrointestinal disorders) | 7 (25)
GASTROINTESTINAL:: Salivary gland changes/saliva (Gastrointestinal disorders) | 1 (7)
GASTROINTESTINAL:: Taste alteration (dysgeusia) (Gastrointestinal disorders) | 5 (16)
GASTROINTESTINAL:: Vomiting (Gastrointestinal disorders) | 2 (2)
HEMORRHAGE/BLEEDING:: Hemorrhage, GI:: Oral cavity (Blood and lymphatic system disorders) | 1 (1)
HEMORRHAGE/BLEEDING:: Hemorrhage, pulmonary/upper respiratory:: Nose (Blood and lymphatic system disorders) | 1 (1)
METABOLIC/LABORATORY:: ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 1 (2)
METABOLIC/LABORATORY:: AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 1 (2)
METABOLIC/LABORATORY:: Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 3 (4)
METABOLIC/LABORATORY:: Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1 (1)
METABOLIC/LABORATORY:: CPK (creatine phosphokinase) (Metabolism and nutrition disorders) | 2 (2)
METABOLIC/LABORATORY:: Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 (1)
METABOLIC/LABORATORY:: Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 2 (3)
METABOLIC/LABORATORY:: Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 4 (7)
METABOLIC/LABORATORY:: Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1 (1)
METABOLIC/LABORATORY:: Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 2 (5)
METABOLIC/LABORATORY:: Metabolic/Laboratory - Other (Specify, __) (Metabolism and nutrition disorders) | 1 (1) — High LDH
METABOLIC/LABORATORY:: Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 2 (2)
METABOLIC/LABORATORY:: Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (1)
METABOLIC/LABORATORY:: Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 (2)
METABOLIC/LABORATORY:: Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (2)
METABOLIC/LABORATORY:: Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 3 (4)
MUSCULOSKELETAL/SOFT TISSUE:: Extremity-upper (function) (Musculoskeletal and connective tissue disorders) | 1 (1)
NEUROLOGY:: Ataxia (incoordination) (Nervous system disorders) | 1 (1)
NEUROLOGY:: Cognitive disturbance (Nervous system disorders) | 1 (1)
NEUROLOGY:: Dizziness (Nervous system disorders) | 5 (5)
NEUROLOGY:: Neurology - Other (Specify, __) (Nervous system disorders) | 1 (1) — Dizziness
PAIN:: Pain:: Abdomen NOS (Musculoskeletal and connective tissue disorders) | 2 (8)
PAIN:: Pain:: Back (Musculoskeletal and connective tissue disorders) | 1 (5)
PAIN:: Pain:: Bone (Musculoskeletal and connective tissue disorders) | 1 (21)
PAIN:: Pain:: Chest wall (Musculoskeletal and connective tissue disorders) | 1 (2)
PAIN:: Pain:: Extremity-limb (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN:: Pain:: Head/headache (Nervous system disorders) | 5 (8)
PAIN:: Pain:: Muscle (Musculoskeletal and connective tissue disorders) | 3 (4)
PAIN:: Pain:: Neck (Musculoskeletal and connective tissue disorders) | 1 (5)
PAIN:: Pain:: Pain NOS (Nervous system disorders) | 1 (1)
PAIN:: Pain:: Pelvis (Musculoskeletal and connective tissue disorders) | 1 (4)
PULMONARY/UPPER RESPIRATORY:: Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
PULMONARY/UPPER RESPIRATORY:: Fistula, pulmonary/upper respiratory:: Lung (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY/UPPER RESPIRATORY:: Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 1 (1) — nasal drying

LIMITATIONS AND CAVEATS:
Study did not meet accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No